CLINICAL TRIAL: NCT00003592
Title: Phase III Randomized Trial of Methotrexate vs. Paclitaxel in Cisplatin-Ineligible Patients With Advanced Squamous Cell Carcinoma of the Head and Neck
Brief Title: Methotrexate Compared With Paclitaxel in Treating Patients With Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066662; E-7397
Record Dates: First submitted 1999-11-01; First posted 2004-06-16 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Head and Neck Cancer
Keywords: stage IV salivary gland cancer; recurrent salivary gland cancer; salivary gland squamous cell carcinoma; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Methotrexate; Paclitaxel

INTERVENTIONS:
Drug: methotrexate
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether methotrexate or paclitaxel is more effective in treating patients with advanced head and neck cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of methotrexate with that of paclitaxel in treating patients who have advanced head and neck cancer that cannot be treated with cisplatin.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the progression free survival, median survival, and overall survival in cisplatin-ineligible patients with advanced squamous cell carcinoma of the head and neck following weekly outpatient methotrexate (arm I) versus paclitaxel (arm II). II. Compare the response rate of patients in the two treatment arms. III. Compare the Trial Outcome Index scores of patients in the two treatment arms. IV. Compare the weight change, neurologic toxicity, and mucositis scores of patients in the two treatment arms.

OUTLINE: This is a randomized study. Patients are stratified by performance status (0-1 vs 2) and age (less than 60 vs at least 60). Patients are randomized to receive methotrexate IV bolus every week for 4 weeks (arm I) or paclitaxel IV over 1 hour every week for 4 weeks (arm II). All patients receive at least 4 weeks of treatment (1 course). Patients continue treatment for a total of 6 courses in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months for 2 years, every 6 months for 3 years, and annually thereafter.

PROJECTED ACCRUAL: There will be 230 patients accrued into this study over 2.4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed advanced, incurable, squamous cell carcinoma of the head and neck Recurrent disease in a previously irradiated field must be biopsy proven or documented unequivocally by physical exam or radiograph(s) Measurable or evaluable disease Patients with ECOG performance status of 0-1 must be ineligible for protocol E-1395 and unable to tolerate cisplatin-based therapy for 1 or more of the following reasons: Hearing loss that precludes cisplatin Unable to handle a fluid load necessitated by cisplatin-based treatment, due to underlying cardiac or pulmonary disease Mild renal insufficiency (creatinine 1.6-2.0 mg/dL) or creatinine clearance of 40-60 mL/min that would make cisplatin treatment difficult, if not dangerous History of brain metastases allowed if disease has stabilized or improved after radiation and/or craniotomy No history of carcinomatous meningitis

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 (See Disease Characteristics) Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,800/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT and SGPT no greater than 5 times upper limit of normal Renal: See Disease Characteristics Creatinine no greater than 2.0 mg/dL No evidence of symptomatic hypercalcemia Cardiovascular: See Disease Characteristics No active angina or uncontrolled arrhythmias Metabolic: No uncontrolled diabetes; no random blood sugar at least 300 mg/dL Neurological: No evidence of ongoing grade 2 or greater peripheral sensory neuropathy Pulmonary: See Disease Characteristics Other: No other concurrent, active, invasive malignancies No significant detectable infection Not pregnant or nursing Effective contraception required of all fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy except in the adjuvant, neoadjuvant, or radiosensitizing setting No prior chemotherapy for recurrent or persistent disease after definitive local therapy At least 6 months since prior methotrexate or paclitaxel Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics At least 4 weeks since prior radiotherapy Surgery: See Disease Characteristics Recovered from prior surgery

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 1999-04-22 (Actual); Primary Completion 2000-08 (Actual); Study Completion 2004-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey J. Langer, MD, Study Chair — Fox Chase Cancer Center
Locations (20):
- United States (19):
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Lakeside), Chicago, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - University of Rochester Cancer Center, Rochester, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - Ireland Cancer Center, Cleveland, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Veterans Affairs Medical Center - Nashville, Nashville, Tennessee
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
- Pretoria Academic Hospital, Pretoria, South Africa